CLINICAL TRIAL: NCT02267863
Title: A Phase Ia/b Dose Escalation and Expansion, Multicenter, Open-label, Safety, Pharmacokinetic and Pharmacodynamic Study of APTO-253 in Patients With Relapsed or Refractory Acute Myelogenous Leukemia or High-Risk Myelodysplasia
Brief Title: A Study of APTO-253 in Patients With Relapsed or Refractory AML or MDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug manufacturing process and procedure review
Sponsor: Aptose Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 253-HEM1-01
Record Dates: First submitted 2014-10-03; First posted 2014-10-20 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Acute Myelogenous Leukemia in Relapse; Acute Myelogenous Leukemia, Relapsed, Adult; Acute Myelogenous Leukemia, Adult; Acute Myelogenous Leukemia; High Risk Myelodysplasia
Keywords: AML; MDS; Leukemia; Acute Myeloid Leukemia; Aptose; APTO-253; Kinase Inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia | interventions — APTO-253

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation and Expansion (Experimental): APTO-253 will be given in ascending doses in patients with relapsed or refractory AML or high risk MDS (escalation cohort), until the maximum tolerated dose or recommended dose is reached. Followed by up to 30 patients enrolled in the expansion cohort at the recommended dose.
  Interventions: Drug: APTO-253

INTERVENTIONS:
Drug: APTO-253 — APTO-253 will be given in ascending doses starting at 20 mg/m2 until the maximum tolerated dose or recommended dose is reached.

SUMMARY:
This study is being done to evaluate the safety and effectiveness of APTO-253 for the treatment of patients with the condition of acute myelogenous leukemia (AML) or myelodysplastic syndrome (MDS) for which either the standard treatment has failed, is no longer effective, or can no longer be administered safely or poses a risk for your general well being.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase Ia/b dose escalation study of safety, pharmacodynamics, and pharmacokinetics of APTO-253 in ascending cohorts (3+3 design) to determine the MTD or recommended dose in patients with relapsed or refractory acute myelogenous leukemia (AML) or high-risk MDS patients. This is to be followed by a cohort expansion phase at the MTD or recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Life expectancy of at least 2 months
* Off previous cancer therapy for at least 14 days, or 5 half-lives for noncytotoxic agents prior to first study treatment administration
* Patients must have a calculated creatinine clearance >60 mL/min
* Acceptable hematologic, renal and liver functions and coagulation status parameters

Exclusion Criteria:

* Patients with GVHD requiring systemic immunosuppressive therapy
* Uncontrolled leptomeningeal disease, auto-immune hemolytic anemia and uncontrolled and clinical significant disease related metabolic disorder
* Clinically significant intravascular coagulation
* Treatment with other investigational drugs within 14 days prior to first study treatment administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-10; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events of APTO-253 | Cycle 1 (28 days)
  To determine the safety and tolerability of APTO-253 by assessing treatment-related adverse events as assessed by CTCAE v4.0.
Maximum tolerated dose and dose limiting toxicities | Cycle 1 (28 days)
  To determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of APTO-253 when given on days 1, 8, 15, and 22 of each 28-day cycle.
Establish recommended dose for future development of APTO-253 | Up to 7 months
  To establish the dose of APTO-253 recommended for future development of APTO-253 for patients with specific types of hematologic malignancies.

SECONDARY OUTCOMES:
Pharmacokinetic variables including maximum plasma concentration (Cmax) | Cycle 1 (28 days)
  Pharmacokinetic variables including maximum plasma concentration (Cmax)
Pharmacokinetic variables including minimum plasma concentration (Cmin) | Cycle 1 (28 days)
  Pharmacokinetic variables including minimum plasma concentration (Cmin)
Pharmacokinetic variables including Area Under the Curve (AUC) | Cycle 1 (28 days)
  Pharmacokinetic variables including Area Under the Curve (AUC)
Pharmacokinetic variables including volume of distribution | Cycle 1 (28 days)
  Pharmacokinetic variables including volume of distribution
Pharmacokinetic variables including clearance | Cycle 1 (28 days)
  Pharmacokinetic variables including clearance
Pharmacokinetic variables including serum half-life | Cycle 1 (28 days)
  Pharmacokinetic variables including serum half-life
Assess for any evidence of antitumor activity of APTO-253 by hematologic and bone marrow evaluations in acute leukemia and MDS. | Average 2 Cycles (8 weeks)
  To observe patients for any evidence of antitumor activity of APTO-253 by hematologic and bone marrow evaluations in acute leukemia and MDS.
Determine the ability of APTO-253 to alter the expression of pharmacodynamic biomarkers of drug effect. | Average 2 Cycles (8 weeks)
  To determine the ability of APTO-253 to alter the expression of pharmacodynamic biomarkers of drug effect.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Bejar, MD., PhD., Study Director — Aptose Biosciences Inc.
Locations (13):
- United States (13):
  - University of Arizona Cancer Center, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California, Irvine, Orange, California
  - Emory University; Winship Cancer Institute, Atlanta, Georgia
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - University of Rochester; Wilmot Cancer Institute Clinical Trials Office, Rochester, New York
  - University Hospital, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Prisma Health, Institute for Translational Oncology Research, Greenville, South Carolina
  - Baylor Research Institute, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Aptose Biosciences — https://www.aptose.com/clinical-trials/apto-253